CLINICAL TRIAL: NCT02686476
Title: Effect of Empagliflozin on Liver Fat Content in Patients With Type 2 Diabetes: A 12-week Randomized Clinical Study
Brief Title: Effect of Empagliflozin on Liver Fat Content in Patients With Type 2 Diabetes
Acronym: E-LIFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medanta, The Medicity, India (Other)
Responsible Party: Principal Investigator, Dr Mohammad Shafi Kuchay, Endocrinologist, Medanta, The Medicity, India
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMELIFT01
Record Dates: First submitted 2016-02-10; First posted 2016-02-19 (Estimated); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Non Alcoholic Fatty Liver Disease
Keywords: Empagliflozin, Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — empagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Empagliflozin dose group (Active Comparator): Patient Receive Standard of Care with Empagliflozen
  Interventions: Drug: Empagliflozin
- Standard dose group (No Intervention): Standard care for Type 2 Diabetes Mellitus upgraded without Empagliflozin

INTERVENTIONS:
Drug: Empagliflozin — group I (n = 50): T2DM patients receiving standard care for T2DM (metformin, sulfonylurea, DPP-4 inhibitor or insulin, in any combination) plus 10 mg of Empagliflozin per day
  Other Names: Jardiance
  Arms: Empagliflozin dose group

SUMMARY:
Fatty liver disease is an increasingly recognized health problem in patients with type 2 diabetes mellitus (T2DM). Sodium glucose co-transporter type 2 (SGLT-2) inhibitors are a new class of anti-diabetic agents that cause weight loss by inducing glycosuria. The effect of SGLT-2 inhibitors on liver fat content is not evaluated. Empagliflozin is an orally active, selective inhibitor of SGLT-2. We hypothesized that Empagliflozin, when added to standard care for T2DM, would improve fatty liver disease. Therefore, the present study is planned to evaluate the effect of Empagliflozin on the liver fat content.

DETAILED DESCRIPTION:
Fatty liver disease is an increasingly recognized health problem in patients with type 2 diabetes mellitus (T2DM). Sodium glucose co-transporter type 2 (SGLT-2) inhibitors are a new class of anti-diabetic agents that cause weight loss by inducing glycosuria. The effect of SGLT-2 inhibitors on liver fat content is not evaluated. Empagliflozin is an orally active, selective inhibitor of SGLT-2. We hypothesized that Empagliflozin, when added to standard care for T2DM, would improve fatty liver disease. Therefore, the present study is planned to evaluate the effect of Empagliflozin on the liver fat content.

Review of literature

Empagliflozin is a selective SGLT-2 inhibitor, recently approved by the U.S. FDA for use in patients with T2DM. Empagliflozin in patients with type 2 diabetes provided sustained glycemic control and weight loss over 90 weeks and was generally well tolerated (1). Another study demonstrated that Empagliflozin in patients with T2DM resulted in reductions in HbA1c and fasting plasma glucose (FPG), and reductions in body weight compared with placebo. Empagliflozin was well tolerated with a favorable safety profile (2). Some congeners of this class of molecules have been seen to reduce liver fat content in rat models. However, the effect of this drug on liver fat content in humans has not been evaluated.

Research question

Does Empagliflozin reduce liver fat content in patients with T2DM and fatty liver disease?

Aim of the study

To study the effect of Empagliflozin on liver fat content in patients with T2DM

Primary objective

1. To evaluate the change in liver fat content from baseline at week 12

   Secondary objective
2. To evaluate the changes from baseline in pancreatic fat content, visceral fat and subcutaneous fat content at 12 weeks

Material and Methods

Ethical considerations

The trial protocol will be submitted to Medanta ethics committees for approval. The trial will be conducted in accordance with the principles of the Declaration of Helsinki and Good Clinical Practice guidelines. All the patients will be provided with written informed consent before participation.

Patients and study area A total of 100 patients will be enrolled for the study. Consecutive patients attending outpatient Department of Endocrinology and Diabetes for management of diabetes will be enrolled.

Sample Size Calculation:

Assumptions: Change in liver fat content from baseline to week 12 in Empagliflozin dose group (m1) = 6.0 unit Change in liver fat content from baseline to week 12 in Standard dose group (m2) = 10.0 unit

Confidence level -95%, Power - 80%, Coefficient of variation = 80% Formula for sample size calculation: n = (Zα+Zβ)2 * (σ12 + σ22)) / (m1-m2)2, where Zα is the value of normal distribution corresponding to desired confidence level, Zβ is the value of the Normal distribution corresponding to desired power, σ1 and σ2 are the standard deviation of the two groups. With these assumptions the sample size per group works out as 50.

Randomization

SPSS software will be used to generate 100 random numbers between 000 to 999. The random numbers will be divided by 2 and the reminder noted. The reminders 0, & 1 will correspond to Empagliflozin dose and standard dose group respectively. It will be ensured that these are equal in number.

Opaque envelopes will be prepared with serial number on the top and the assigned group inside the envelope.

After recruiting the subjects the envelop with corresponding serial number will be opened and the subjects assign to the relevant groups.

Statistical Analysis Plan:

The analysis will include profiling of patients on different demographic, clinical and laboratory parameters etc. Quantitative data will be presented in terms of means and standard deviation and qualitative/categorical data will be presented as absolute numbers and proportions. Cross tabulation will be generated and chi square test will be used for testing of association. Student t test will be used for comparison of quantitative outcome parameters and standard normal deviate test for proportions. P-value < 0.05 is considered statistically significant. SPSS software will be used for analysis.

All patients will be randomized to one of the following intervention groups: group I (n = 50): T2DM patients receiving standard care for T2DM (metformin, sulfonylurea, DPP-4 inhibitor or insulin, in any combination) plus 10 mg of Empagliflozin per day and group II (n = 50): Standard care for T2DM upgraded without Empagliflozin.

Liver fat content, pancreatic fat content, visceral and subcutaneous fat content will be assessed by magnetic resonance imaging (MRI) proton density fat Fraction (PDFF) at the beginning of study and again after 12 weeks of intervention. PDFF is emerging as a leading MR-based biomarker for noninvasive quantification of hepatic steatosis (3, 4). Multiple human studies have shown that this method accurately estimates PDFF in the liver. Based on these results, this magnitude-based PDFF estimation method now is being used to quantify liver fat in clinical practice in several institutions in the United States and is being used as a biomarker of drug efficacy and drug toxicity by the National Institutes of Health (NIH) and industry in clinical trials (5, 6). This method has been shown to be both accurate, and reproducible (7).

Fatty liver will also be assessed by ultrasonography of liver at the beginning of study and again after 12 weeks of intervention. On ultrasonography, severity of fatty liver will be quantitated using a scoring system (0 = no fatty liver, 1 = mild fatty liver, 2 = moderate fatty liver and 3 = severe fatty liver). Automated body composition analyzer (BCA) will also be used to assess body composition at 0 and 12 weeks.

Laboratory workup Biochemical parameters will include fasting and post-prandial plasma glucose, glycosylated hemoglobin (HbA1C), lipid profile, hemogram, kidney function test (urea, creatinine) and liver function test (total and fractionated bilirubin, alanine transaminase (ALT), aspartate aminotransferase (AST), gamma-glutamyl transpeptidase (GGT), total protein, albumin) before and after the intervention period.

The primary end point

1. Change in liver fat content from baseline at week 12 The secondary end points
2. Change in pancreatic fat content, visceral fat and subcutaneous fat content from baseline at week 12

Confidentiality Precautions will be taken to ensure confidentiality. Data collection forms will not reveal the name of the patients included in study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with T2DM of age 40 years and above
* Fatty liver disease (grade I or more on USG)
* Glycated A1C more than 7.0% but less than 10.0%
* Patient on standard care of T2DM (metformin, sulfonylureas, DPP-4 inhibitors or insulin, in any combination).

Exclusion Criteria:

1. Serum creatinine more than 1.5 mg/dL
2. Pregnancy
3. Participants treated with pioglitazone or vitamin E in the immediate past 6 months
4. Presence of major contraindications to magnetic resonance imaging (cardiac pacemakers, claustrophobia, foreign bodies and implanted medical devices with ferromagnetic properties).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in Liver Fat | 3 Months
  To evaluate the change in liver fat content at baseline and 3 Months

SECONDARY OUTCOMES:
Pancreatic fat content | 3 Months
  To evaluate the changes in pancreatic fat content at baseline and 3 Months
visceral fat | 3 Months
  To evaluate the changes in visceral fat content at baseline and 3 Months
subcutaneous fat | 3 Months
  To evaluate the changes in subcutaneous fat content at baseline and 3 Months

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad S Kuchay, MD,DM, Principal Investigator — Endocrinologist
Locations (1):
- Division Of Endocrinology , Medanta The Medicity Sec 38, Gurgaon, Haryana, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Reeder SB, Cruite I, Hamilton G, Sirlin CB. Quantitative Assessment of Liver Fat with Magnetic Resonance Imaging and Spectroscopy. J Magn Reson Imaging. 2011 Oct;34(4):729-749. doi: 10.1002/jmri.22775. Epub 2011 Sep 16. PMID 22025886
- [Result] Ferrannini E, Seman L, Seewaldt-Becker E, Hantel S, Pinnetti S, Woerle HJ. A Phase IIb, randomized, placebo-controlled study of the SGLT2 inhibitor empagliflozin in patients with type 2 diabetes. Diabetes Obes Metab. 2013 Aug;15(8):721-8. doi: 10.1111/dom.12081. Epub 2013 Mar 4. PMID 23398530
- [Result] Rosenstock J, Seman LJ, Jelaska A, Hantel S, Pinnetti S, Hach T, Woerle HJ. Efficacy and safety of empagliflozin, a sodium glucose cotransporter 2 (SGLT2) inhibitor, as add-on to metformin in type 2 diabetes with mild hyperglycaemia. Diabetes Obes Metab. 2013 Dec;15(12):1154-60. doi: 10.1111/dom.12185. Epub 2013 Aug 22. PMID 23906374
- [Result] Reeder SB, Sirlin CB. Quantification of liver fat with magnetic resonance imaging. Magn Reson Imaging Clin N Am. 2010 Aug;18(3):337-57, ix. doi: 10.1016/j.mric.2010.08.013. PMID 21094444
- [Result] Le TA, Chen J, Changchien C, Peterson MR, Kono Y, Patton H, Cohen BL, Brenner D, Sirlin C, Loomba R; San Diego Integrated NAFLD Research Consortium (SINC). Effect of colesevelam on liver fat quantified by magnetic resonance in nonalcoholic steatohepatitis: a randomized controlled trial. Hepatology. 2012 Sep;56(3):922-32. doi: 10.1002/hep.25731. Epub 2012 Jul 2. PMID 22431131
- [Result] Krishan S, Jain D, Bathina Y, Kale A, Saraf N, Saigal S, Choudhary N, Baijal SS, Soin A. Non-invasive quantification of hepatic steatosis in living, related liver donors using dual-echo Dixon imaging and single-voxel proton spectroscopy. Clin Radiol. 2016 Jan;71(1):58-63. doi: 10.1016/j.crad.2015.10.002. Epub 2015 Nov 7. PMID 26555703
- [Derived] Kuchay MS, Krishan S, Mishra SK, Farooqui KJ, Singh MK, Wasir JS, Bansal B, Kaur P, Jevalikar G, Gill HK, Choudhary NS, Mithal A. Effect of Empagliflozin on Liver Fat in Patients With Type 2 Diabetes and Nonalcoholic Fatty Liver Disease: A Randomized Controlled Trial (E-LIFT Trial). Diabetes Care. 2018 Aug;41(8):1801-1808. doi: 10.2337/dc18-0165. Epub 2018 Jun 12. PMID 29895557